CLINICAL TRIAL: NCT06215950
Title: A Phase I Clinical Study to Assess the Safety and Efficacy of CD70-targeted CAR-T in the Treatment of CD70-positive Advanced/Metastatic Gynecologic Cancer
Brief Title: A Clinical Research About CD70-targeted CAR-T in the Treatment of CD70-positive Advanced/Metastatic Gynecologic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC061
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Cervix Cancer; Metastatic Cancer; Advanced Cancer; Gynecologic Cancer
Keywords: CAR-T; CD70
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD70 CAR-T cells
- intraperitoneal injection of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD70 CAR-T cells

INTERVENTIONS:
Biological: CD70 CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were transfused intravenically
  Arms: Intravenous of CD70-targeted CAR-T
Biological: CD70 CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were injected intraperitoneally
  Arms: intraperitoneal injection of CD70-targeted CAR-T

SUMMARY:
This is a single-center, double-arm, open-label study. this study plans to evaluate the safety and efficacy of CD70-targeting CAR-T cells in the treatment of CD70-positive advanced/metastatic Gynecologic Cancer, and obtain recommended doses and infusion patterns.

DETAILED DESCRIPTION:
The research designs to follow 2 groups：Intravenous infusion group and Intraperitoneal injection group；each group sets up 2 phases,the first phase is dose discovery phase to obtain recommended doses,the second phase is dose expansion phase to verify the safety in the recommended doses. In the discovery phase,each group puts up 4 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 12 subjects with CD70-positive advanced/metastatic solid tumors.In the dose expansion phase,each group will choose one or two dose groups to verify the safety and efficacy at this dose,and plan to recruit about 6 subjects in each dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Advanced/metastatic gynecological tumor confirmed by histopathology or cytology (paraffin sections or fresh biopsy tumor tissue specimens) (CD70 positive tumor expression (CD70 positive tumor confirmed by histology or pathology (IHC 3+));
3. Failure or intolerance after standard treatment (disease progression or intolerance such as surgery, chemotherapy, radiotherapy, targeted therapy, etc.), and currently no effective treatment;
4. According to the RECIST version 1.1 standard, there is at least one measurable diameter and evaluable target lesion. Measurable lesions are defined as: extranodal lesions with CT scan diameter ≥10mm, lymph node lesions with CT scan diameter ≥15mm, scan layer thickness ≤ 5mm, and have not received local treatment;
5. ECOG 0 ~ 2 points ;
6. Expected survival time is more than 12 weeks;
7. No serious mental disorders;
8. The functions of important organs are basically normal:

   1. Hematopoietic function: neutral granules >1.0×109/L, platelet >75×109/L, hemoglobin >80g/L;
   2. Cardiac function: Echocardiography indicated cardiac ejection fraction ≥50%, and no obvious abnormality was found in electrocardiogram;
   3. Renal function: serum creatinine ≤2.0×ULN;
   4. Liver function: ALT and AST ≤2.0×ULN (patients with liver tumor infiltration can be relaxed to ≤3.0×ULN);
   5. Total bilirubin ≤2.0×ULN (Gilbert syndrome or liver tumor infiltration can be relaxed to ≤3.0×ULN);
   6. Blood oxygen saturation in non-oxygen state>92%.
9. Have the criteria for simple or intravenous blood collection, and no other contraindications for cell collection;
10. The subject agrees to use a reliable and effective contraceptive method for contraception (excluding safe period contraception) within 1 year from signing the informed consent to receiving the CAR T cell infusion;
11. The subject or his/her guardian agrees to participate in the clinical trial and signs the ICF, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Received anti-CD70 drug therapy before screening;
2. Active/symptomatic central nervous system metastasis or meningeal metastasis at the time of screening; Treated subjects with brain metastases can only be enrolled if no radiographically demonstrated progression is demonstrated ≥4 weeks after the end of treatment.
3. Received any of the following treatments prior to screening:

   1. Participated in other interventional clinical studies before screening, including: the time of last use of unmarketed new drugs less than 3 months from cell transfusion, or the time of last use of marketed drugs less than 5 half-lives from cell transfusion;
   2. Received anti-tumor therapy such as chemotherapy or targeted therapy within 2 weeks of preapheresis or at least 5 half-lives (whichever is shorter); Received systemic radiation within 4 weeks and local radiation within 2 weeks; Or received radioactive drugs (strontium, samarium) within 8 weeks prior to treatment.
   3. Systemic corticosteroid therapy with doses greater than 10mg/ day of prednisone (or equivalent doses of other corticosteroids) within 2 weeks of preapheresis (in the absence of active autoimmune disease, inhaled or topical steroid use and adrenocortical replacement with doses greater than 10mg/ day of prednisone efficacy dose are permitted);
   4. Received live attenuated vaccine within 4 weeks prior to screening;
4. There is an active or uncontrolled infection requiring systemic treatment within 1 week prior to screening;
5. Had malignancies other than the target tumor within 3 years prior to screening, except for malignancies that had received radical treatment and had no known active disease for ≥3 years prior to enrollment; Or adequately treated non-melanoma skin cancer with no evidence of disease;
6. Have any of the following heart conditions:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Had myocardial infarction or coronary artery bypass grafting (CABG) within ≤6 months before enrollment;
   3. A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy.
7. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc.
8. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal range; Positive for human immunodeficiency virus (HIV) antibodies; Syphilis positive; Cytomegalovirus (CMV) DNA test positive;
9. The subject has a history of venous embolism (e.g., pulmonary embolism) and currently requires anticoagulant therapy, or if: a. Bleeding with grade 3 to 4 persists for more than 30 days; b. have sequelae from venous embolism (e.g. persistent dyspnea and hypoxia); (Note: Participants who have venous embolism but do not meet the above criteria can participate in the test);
10. Poorly controlled hypertension, defined as systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥90mmHg (Blood pressure values are measured based on the average of 3 readings at least 2 minutes apart, patients with blood pressure ≥150/90 MMHG at initial screening may receive antihypertensive treatment, if well controlled after treatment, And blood pressure < 150/90mmHg can be screened);
11. Women who are pregnant or breastfeeding, and male or female subjects who plan to have a family within 1 year after receiving CAR T cell transfusion;
12. Conditions deemed unsuitable for participation in the study by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CD70 CAR-T cells infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of CD70 CAR-T cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Disease control rate of CAR-T cell preparations in CD70 positive advanced malignancies [Effectiveness] | 3 months
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Objective response rate (ORR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 3 months
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CD70-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CD70-CAR-T cell infusion to death from any cause (Assessed based on RECIST criteria)
AUCS of CD70 CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CD70 CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CD70 CAR-T cells expanded in peripheral blood
TMAX of CD70 CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CD70 CAR-T cells[Cell dynamics] | 3 months
  Concentration levels of CAR-T-related serum cytokines such as CRP, IL-6, ferritin at each time point，which measured by Chemiluminescence method

OTHER OUTCOMES:
The correlation between CD70 positive rate and safety | 2 years
  assessment the correlation between CD70 positive rate and the incidence of CRA and ICANS
Correlation between CD70 positive rate and efficacy | 2 years
  assessment the correlation between CD70 positive rate and the disease control rate，Disease control rate: including CR, PR and SD
Overall survival(OS)of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CD70-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)
Progress-free survival(PFS) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CD70-CAR-T cell infusion to death from any cause or the first assessment of progression (Assessed by investigators based on IRECIST criteria)
Duration of Response (DOR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Guantai Ni, M.D, Principal Investigator — First Affiliated Hospital of Wannan Medical College
Locations (1):
- The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No